CLINICAL TRIAL: NCT03199690
Title: Phase One, Open Lab Study to Investigate the Impact of Rifampicin Administration on the PK of Dolutegravir When Dosed Once Daily at 50 or 100 mg in Healthy Volunteers
Brief Title: A Clinical Study Investigating Rifampicin and Dolutegravir in Combination in Healthy Volunteers
Acronym: RADIO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Stephens Clinical Research (Other)
Responsible Party: Sponsor
Organization: St Stephens Aids Trust (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SSCR103
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: HIV-1-infection; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — dolutegravir; Rifampin

STUDY DESIGN:
Intervention Model Description: open label, single centre, sequential pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Single arm trial design based on the dosing regimen below:
  Day 1 - 7
  - Dolutegravir 50 mg once daily with food
  Day 8 - 14 - Dolutegravir 100 mg once daily with food
  Day 15 - 28
  - Rifampicin 600 mg once daily
  Day 29 - 35 - Rifampicin 600 mg once daily & Dolutegravir 50 mg once daily
  Day 36 - 42
  - Rifampicin 600 mg once daily & Dolutegravir 100 mg once daily
  Interventions: Drug: Dolutegravir; Drug: Rifampicin

INTERVENTIONS:
Drug: Dolutegravir — Antiviral (integrase inhibitor)
  Other Names: Tivicay
Drug: Rifampicin — Antibiotic
  Other Names: Rifidan

SUMMARY:
The purpose of the study is to see how the drug Dolutegravir is broken down by your body, when taken with another drug called Rifampicin. Dolutegravir is given to people as a treatment for HIV. Rifampicin is given to people as a treatment for tuberculosis.

DETAILED DESCRIPTION:
The integrase inhibitor under investigation in this study, Dolutegravir (DTG), is relatively new to the market only having been approved in 2014. DTG is now being used on a large scale to treat HIV-1 positive patients, therefore robust drug-drug interaction data is required for medications that are prescribed with DTG.

Tuberculosis is biggest killer of patients that are co-infected with the HIV-1 virus, killing over 25% of the population. There is an unmet need for data concerning DTG once daily dosing in the presence of rifampicin (RIF), the widely used anti-tuberculosis antibiotic. This is the main purpose of this investigative study.

The design of the study is an open label, single site pharmacokinetic (PK) study to measure the blood plasma concentration of DTG in the presence of RIF.

The study will recruit 18-63 years old healthy volunteers, either male or non-pregnant females. Subjects will be recruited at the single study site. A site in the United Kingdom will be selected based on its past experience in the HIV field, and its ability to recruit 16 subjects from their healthy volunteer database.

The study period is expected to be 43 days, excluding screening and follow-up. The most significant procedures in terms of study data will be pharmacokinetic (PK) sampling days 7, 14, 35 and 42. On these days PK sampling will occur over a 24 hour period, mapping out the blood concentrations of DTG in the presence of RIF.

There will also be a pharmacogenomic sub-study included in the study design. Researchers have included this because the HIV investigator community agrees that a pharmacogenomic approach to HIV treatment is important to understand why patients show different degrees of virological responses or drug toxicity.

This research is funded by Wits Health Consortium, and sponsored by St Stephens Clinical Research.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females.
3. Between 18 to 60 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive (with weight ≥50kg).
5. Alanine aminotransferase, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
6. Women of childbearing potential (WOCBP - definition in Appendix 4) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 3 months after the study.

   A female may be eligible to enter and participate in the study if she:
   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
   3. True abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 4 weeks after discontinuation of all study medications. (When this is in line with the preferred and usual lifestyle of the subject.) (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), and withdrawal are not acceptable methods of contraception].
   4. Any non-hormonal intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see protocol appendix 4 for an example listing of approved IUDs);
   5. Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject; Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of IP.
7. Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 4 must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study (see inclusion criteria 6);

   * True abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 4 weeks after discontinuation of all study medications (When this is in line with the preferred and usual lifestyle of the subject.) (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), and withdrawal are not acceptable methods of contraception].
   * Any non-hormonal intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 4 for an example listing of approved IUDs);
   * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject; Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP.
8. Willing to consent to their personal details being entered onto the TOPS database
9. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
10. Registered with a GP in the UK

Exclusion Criteria:

1. Any clinically significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen or C antibody
4. Positive blood screen for HIV-1 or 2 by antibody/antigen assay
5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
6. Current or recent (within three months) gastrointestinal disease.
7. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
8. Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within three months of first dose of study drug
9. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
10. Females of childbearing potential without the use of effective birth control methods, or not willing to continue practising these birth control methods for at least 4 weeks after the end of the treatment period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
To investigate the pharmacokinetics of DTG 50 or 100 mg OD in the presence of RIF 600 mg OD in healthy volunteers as measured by trough concentration (Ctrough) | 43 days
  Ctrough is defined as the concentration at 24 hours after the observed drug dose.
To investigate the pharmacokinetics of DTG 50 or 100 mg OD in the presence of RIF 600 mg OD in healthy volunteers as measured by maximum observed plasma concentration (Cmax) | 43 days
  Maximum observed plasma concentration (Cmax).
To investigate the pharmacokinetics of DTG 50 or 100 mg OD in the presence of RIF 600 mg OD in healthy volunteers as measured by elimination half-life (t1/2) | 43 days
  Elimination half-life (t1/2)
To investigate the pharmacokinetics of DTG 50 or 100 mg OD in the presence of RIF 600 mg OD in healthy volunteers as measured by time point at Cmax (Tmax) | 43 days
  Time point at Cmax (Tmax)
To investigate the pharmacokinetics of DTG 50 or 100 mg OD in the presence of RIF 600 mg OD in healthy volunteers as measured by total drug exposure. | 43 days
  Total drug exposure, expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h).

IPD SHARING:
Plan to Share IPD: No